CLINICAL TRIAL: NCT01489215
Title: Interventions for Sleep Problems in Early Childhood:The Role of Child, Parental and Intervention Factors
Brief Title: Interventions for Sleep Problems in Early Childhood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Israel Science Foundation (Other); U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TASMC-11-YS-0522-CTIL
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Presenteeism; Banking, Personal

ARMS (3):
- Clinical group-"presence" intervention (Experimental): The "Presence" intervention is based on based on the principles of graduated extinction, which has been defined has been defined as "effective and recommended therapy in the treatment of bedtime problems and night wakings" by the Standard of Practice Committee of the American Academy of Sleep Medicine.
  Interventions: Behavioral: "presence"
- Clinical group-"checking" intervention (Experimental): The "Checking" training is based on the principles of graduated extinction, which has been defined has been defined as "effective and recommended therapy in the treatment of bedtime problems and night wakings" by the Standard of Practice Committee of the American Academy of Sleep Medicine
  Interventions: Behavioral: "checking"
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: "presence" — constant presence of the parent in the child's room throughout the night during the first week of the intervention. In addition to sleeping near the child's crib, the parents repeat the same routines as in the "checking" method if the child is actively protesting or crying.
  Arms: Clinical group-"presence" intervention
Behavioral: "checking" — putting the child into the crib at bedtime and leaving the room with repeated quick visits every 5 minutes if the child is actively protesting or crying, providing brief reassurance, helping the child to resume a sleeping position.
  Arms: Clinical group-"checking" intervention

SUMMARY:
This study will inform the field about underlying mechanisms associated with infant sleep problems and will deepen the understanding of the intervention process. The study will provide detailed information on the intervention process itself and will explore how behavioral sleep interventions affect broader infant outcome.

ELIGIBILITY:
Inclusion Criteria:

* infants at age range 9-18 months;
* healthy infants with no significant health problems;
* two-parents families;
* parents who master the Hebrew language.
* significant sleep problem lasting more than 3 months:

Our definition for a significant sleep problem in this age range is based on meeting at least one of the following three criteria for the baseline week:

* an average of three or more night-wakings per night;
* an average wake period of at least 30 minute per night between sleep onset and morning rise time;
* more than 30 minutes to fall asleep each night with protests for attention.

Exclusion Criteria:

* Infants not meeting the inclusion criteria at the baseline assessment will be excluded from the study.

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Improved infant sleep | base line to one month follow-up
  Less parental involvement in falling asleep, less night wakings, heightened sleep efficacy

SECONDARY OUTCOMES:
improvement in infant emotion regulation and in parent-infant interaction | one month follow-up to one year follow-up
  infant heightened ability to regulate emotion when frustrated, a more secure infant attachment to mother, less infant withdrawal and more maternal sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Yakov Sivan, Prof., Principal Investigator — Tel-Aviv Sourasky Medical Center

REFERENCES:
- [Derived] Kahn M, Livne-Karp E, Juda-Hanael M, Omer H, Tikotzky L, Anders TF, Sadeh A. Behavioral interventions for infant sleep problems: the role of parental cry tolerance and sleep-related cognitions. J Clin Sleep Med. 2020 Aug 15;16(8):1275-1283. doi: 10.5664/jcsm.8488. PMID 32279703
- [Derived] Kahn M, Juda-Hanael M, Livne-Karp E, Tikotzky L, Anders TF, Sadeh A. Behavioral interventions for pediatric insomnia: one treatment may not fit all. Sleep. 2020 Apr 15;43(4):zsz268. doi: 10.1093/sleep/zsz268. PMID 31676910